CLINICAL TRIAL: NCT03228056
Title: Postoperative Pain After Single Port, Two Ports and Three Ports Video-assisted Thoracic Surgery Lobectomy in Cancer Patients: A Randomized Controlled Trial
Brief Title: Postoperative Pain After Single Port, Two Ports and Three Ports VATS Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pulmonary Hospital Zakopane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHZakopane
Record Dates: First submitted 2017-06-09; First posted 2017-07-24 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer
Keywords: postoperative pain; videothoracoscopic surgery; thoracic epidural analgesia; lung lobectomy
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- uniportal VATS lobectomy (Experimental): * uniportal VATS lobectomy
  * thoracic epidural block (0.125% bupivacaine with epinephrine 1:50000, continuous infusion 3-4 ml/hour)
  * ketoprofene 100 mg i.v every 12 hours
  * paracetamol 1000 mg i.v every 8 hours
  * rescue doses of morphine in PCA system (bolus dose 2 mg i.v)
  * pain intensity measured in VAS scale
  Interventions: Diagnostic Test: pain intensity measured in VAS scale
- two-ports VATS lobectomy (Active Comparator): * two-ports VATS lobectomy
  * thoracic epidural block (0.125% bupivacaine with epinephrine 1:50000, continuous infusion 3-4 ml/hour)
  * ketoprofene 100 mg i.v every 12 hours
  * paracetamol 1000 mg i.v every 8 hours
  * rescue doses of morphine in PCA system (bolus dose 2 mg i.v)
  * pain intensity measured in VAS scale
  Interventions: Diagnostic Test: pain intensity measured in VAS scale
- three-ports VATS lobectomy (Active Comparator): * three-ports VATS lobectomy
  * thoracic epidural block (0.125% bupivacaine with epinephrine 1:50000, continuous infusion 3-4 ml/hour)
  * ketoprofene 100 mg i.v every 12 hours
  * paracetamol 1000 mg i.v every 8 hours
  * rescue doses of morphine in PCA system (bolus dose 2 mg i.v)
  * pain intensity measured in VAS scale
  Interventions: Diagnostic Test: pain intensity measured in VAS scale

INTERVENTIONS:
Diagnostic Test: pain intensity measured in VAS scale — Pain intensity in 0-100 mm VAS scale is measured every 4 hours on standard ruler beginning from the end of the surgery.

SUMMARY:
This single-center, prospective, randomized controlled trial was designed to assess and compare the postoperative pain after VATS lobectomy performed though one, two and three incisions. The primary outcome measure is pain intensity measured in VAS scale. The secondary outcome measure is cumulative morphine consumption up to 72 hours after surgery

DETAILED DESCRIPTION:
The best VATS technique for lobectomy has not been well defined yet. Most of the authors describe the VATS approach to lobectomy via 2 to even 4 incisions. The final step in the evolution of the technique is the use of a single-port approach. If conventional multiportal VATS is superior to open thoracotomy by virtue of minimizing surgical access trauma, then further reduction in such access trauma should yield even greater benefits. Therefore, reducing the number of wounds from three or four to just one, should, in theory, lead to less pain, paresthesia, and morbidity as well as faster recovery. However, critics of the uniportal VATS approach may raise concerns about whether this most minimally invasive surgical approach for lung surgery may compromise safety and treatment efficacy. In addition, there's the concern about true invasiveness of the procedure. This prospective, randomized controlled trial was designed to compare the postoperative pain after VATS lobectomy performed through one, two and three incisions. The primary outcome measure is pain intensity measured in VAS scale. The secondary outcome measures are cumulative morphine consumption up to 72 hours after surgery in 4-hour intervals and dynamic spirometry (PEF, FEV1 and FVC) measured daily at the bedside up to 72 hours after surgery. All patients will receive the same regimen of postoperative analgesia based on thoracic epidural block, non-steroidal anti-inflammatory drugs and rescue doses of morphine in PCA system. The side effects and complications including atelectasis, pneumonia, atrial fibrillation, urine retention, hypotension, respiratory depression and sedation will be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status 1-3
2. undergo videothoracoscopic lung lobectomy
3. forced expiratory volume in 1 second (FEV1) >1,5 l/min
4. no contraindications for epidural anesthesia
5. ability to comprehend principles of VAS pain examination method and to communicate in accordance with them.

Exclusion Criteria:

1. prior to the study: contraindications for local anesthesia, ASA>3, FEV1<1,5 l/min, conditions disabling the patient from comprehending the principles of VAS pain examination, known allergy to used medications.
2. during the study: failure to place epidural catheter, decision to abandon lobar resection (e.g. in case of neoplastic dissemination), intraoperative conversion to thoracotomy, intraoperative anatomical obstacles to distribution of local anesthetics, conditions disabling the patient from pain evaluation by means of VAS method (e.g. postoperative delirium), necessity to administer other pharmaceuticals influencing pain perception (e.g. sedatives), necessity of mechanical ventilation, interruption of local anesthesia as a result of technical problems (e.g. damage or slippage of catheter).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to 72 hours after the end of surgery
  0-100 mm VAS scale measured every 4 hours on standard ruler beginning from the end of the surgery

SECONDARY OUTCOMES:
opioid consumption | up to 72 hours after the end of surgery
  cumulative rescue morphine consumtion (PCA) in miligrams
rate of complications | up to 72 hours after the end of surgery
  frequency of postoperative complications (atelectasis, pneumonia, atrial fibrillation, urine retention, hypotension, respiatory depression, sedation)

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Zieliński, PhD, Principal Investigator — Pulmonary Hospital, Zakopane, Poland
Locations (2):
- Poland (2):
  - Pulmonary Hospital, Zakopane, Malopolska
  - Pulmonary Hospital, Zakopane

IPD SHARING:
Plan to Share IPD: No